CLINICAL TRIAL: NCT05523141
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of ASC10 Tablets and an Open-label, Crossover Design to Evaluate the Food Effect on PK of ASC10 in Healthy Subjects
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and the Food Effect on PK of ASC10 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASC10-101
Record Dates: First submitted 2022-08-30; First posted 2022-08-31 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: SARS CoV 2 Infection
Keywords: ASC10; RdRp; Healthy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC10 (Experimental): Part 1: Participants will be randomized to receive 100 to 1600 mg ASC10 (including 6 cohorts) in an double-blind manner
  Part 2: Participants will be randomized to receive two single 800 mg doses (fed or fasted)
  Interventions: Drug: ASC10
- Placebo (Placebo Comparator): Part 1: Participants will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASC10 — Part 1:
  Participants will be randomized to receive twice daily dosing either ASC10 or Placebo for 5.5 days, in an double-blind manner
  Part 2:
  Two single oral doses of ASC10 will be administered to participants, in an open-label manner
  Arms: ASC10
Drug: Placebo — Part 1:
  Participants will be randomized to receive twice daily dosing either ASC10 or Placebo, in an double-blind manner
  Arms: Placebo

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled study to evaluate safety, tolerability, and pharmacokinetics of ASC10 tablets and an open-label, crossover design to evaluate the food effect on PK of ASC10 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers between the ages 18 and 45, inclusive
* Those who do not have plans for pregnancy within six months and are willing to take effective contraceptive measures from the first dose of the study drug to 3 months after the last dose.
* If male, agree to use adequate contraception throughout the study and for at least 3 months after the last dose of study drug.
* Body mass index (BMI) was between 19 and 26 kg/m^2. Weight ≥50 kg for males and ≥45 kg for females.

Exclusion Criteria:

* Females who are pregnant, planning to become pregnant, or breastfeeding.
* Has any current or historical disease or disorder of the hematological system or significant liver disease or family history of bleeding/platelet disorders.
* Has a history of cancer (other than basal cell or squamous cell cancer of the skin), rheumatologic disease or blood dyscrasias.
* Has a history of blood dizziness or difficulty in blood collection.
* Has donated blood within 30 days, plasma within 2 weeks, or platelets within 6 weeks before the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Part1: Number of participants with Treatment Emergent Adverse Events (TEAEs) in multiple ascending dose (MAD) | From screening through study completion, up to 12 days
Part1: Number of Participants With Clinically Significant Change From Baseline in Vital Signs in MAD | From screening through study completion, up to 12 days
  Vital signs evaluation includes: systolic and diastolic blood pressure (BP), temperature, respiratory rate and pulse rate.
Part1: Number of Participants With Laboratory Abnormalities in MAD | From screening through study completion, up to 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Yunqing Qiu, Master, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Liu J, Zhao Q, Zhai Y, Wu X, Kai J, Ruan J, Wu M, Wu M, Zhou Z, Yan Y, Wu JJ, Qiu Y. Safety, tolerability and pharmacokinetics of ASC10, a novel oral double prodrug of a broad-spectrum antiviral agent, beta-d-N4-hydroxycytidine: results from a randomized, double-blind, placebo-controlled phase 1 study in Chinese healthy subjects. Expert Opin Investig Drugs. 2024 Aug;33(8):867-876. doi: 10.1080/13543784.2024.2377318. Epub 2024 Jul 12. PMID 38988285